CLINICAL TRIAL: NCT00503061
Title: A Pharmaceopidemiological Study in Patients Who Use Symbicort Turbuhaler as Maintenance and Reliever Therapy (Symbicort SMART) Capturing Over Use and Under Use Via the General Practice Research Database
Brief Title: A Pharmaceopidemiological Study in Patients Who Use Symbicort SMART
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Tomas Andersson, MSD, AstraZeneca Pharmaceuticals
Other Study IDs: D5890C00017; GPRD
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Bronchial Asthma
Keywords: pharmaceopidemiological; Symbicort SMART; GPRD
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
To investigate how common it is that patients using Symibort SMART take high average daily doses that are not considered appropriate by their physician (overuse) or are hospitalised due to their asthma at least partly due to underuse.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosis, patient registered with the prescribing physician for at least one year before the qualifying prescription of Symbicort, prescription of Symbicort SMART after UK launch of the concept

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population comes from Primary Care Clinics and Pulmonary Experts
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2007-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catriona McMahon, MD, Principal Investigator — AZ UK MC; Tomas Andersson, MD, Study Director — AZ R&D Lund
Locations (1):
- Research Site, London, United Kingdom